CLINICAL TRIAL: NCT05014113
Title: A Retrospective Study Evaluating Clinical and Radiographic Early Outcomes of Total Hip Arthroplasty With DELTA ST-C Cup and MINIMA Stem.
Brief Title: H-28 DELTA ST-C and Minima Retrospective Study.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Limacorporate S.p.a (Industry)
Responsible Party: Sponsor
Other Study IDs: H-28
Record Dates: First submitted 2021-08-09; First posted 2021-08-20 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Osteoarthritis, Hip
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: DELTA-ST cup in combination with MINIMA stem — Advance articular destruction generated by primary degenerative or post-traumatic arthrosis or reumatoid arthritis; fracture or avascular necrosis; congenital or acquired deformity.

SUMMARY:
The study aims to assess the clinical and radiographic outcomes of DELTA ST-C in combination with MINIMA stem at 3 years after primary THA surgery, and to evaluate the overall survivorship of the implant.

ELIGIBILITY:
Inclusion Criteria:

* Underwent to a THA with DELTA ST-C cup and MINIMA stem in 2017 onwards
* Both genders
* Any race
* A diagnosis in the target hip of one or more of the following:

  1. Non-inflammatory degenerative joint disease such as osteoarthritis, avascular necrosis
  2. Rheumatoid Arthritis
  3. Post-traumatic arthritis
  4. Fractures of femoral neck
  5. Congenital or acquired deformity
* Patient willingness to participate

Exclusion Criteria:

* Local or systemic infection
* Septicaemia
* Persistent acute or chronic osteomyelitis
* Confirmed nerve or muscle lesion compromising hip joint function
* Vascular or nerve diseases affecting the concerned limb
* Poor bone stock (for example due to osteoporosis) compromising the stability of the implant
* Metabolic disorders which may impair fixation and stability of the implant
* Any concomitant disease and dependence that might affect the implanted prosthesis
* Metal hypersensitivity to implant materials
* Required revision of previous standard femoral stem
* Age < 18 years old
* Any clinically significant pathology based on clinical history that the Investigator feels may affect the study evaluation including, but not limited to:

  1. significant neurological or musculoskeletal disorders or disease that may adversely affect gait and compromise functional recovery
  2. neuromuscular or neurosensory deficit which would limit the ability to assess the performance of the device
  3. known metabolic disorders leading to progressive bone deterioration
* Hip replacement on the contralateral side performed within less than one year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of 95 consecutive patients who underwent to a THA with DELTA ST-C cup in combination with MINIMA stem in 2017 onwards at the Psychiko Clinic and are compliant with all the Inclusion and Exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 95 (Estimated)
Dates: Start 2020-09-15 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Harris Hip Score (HHS) | Pre-operative - Month 36
  Assessment of Harris Hip Score from pre-operative baseline up to 3 years after surgery

SECONDARY OUTCOMES:
Stability assessment of DELTA ST-C cup | At discharge - Month 36
  Radiographic analysis and stability assessment of the DELTA ST-C cup as rate of symptomatic radiolucent lines, loosening, and subsidence ≥ 2 mm from discharge (baseline) up to 3-year follow-up
Stability assessment of MINIMA stem | At discharge - Month 36
  Radiographic analysis and stability assessment of the MINIMA stem as rate of symptomatic radiolucent lines, loosening, and subsidence ≥ 2 mm from discharge (baseline) up to 3-year follow-up
Survival rate of the implant | Month 36
  The survival rate of the implant is expressed by Kaplan-Meier estimator
Safety assessment (adverse events) | Intra-operative - Month 36
  Assessment of any possible adverse device event or device-related complication detected and recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Psychiko Clinic (Athens Medical Group), Athens, Psychiko, Greece